CLINICAL TRIAL: NCT03910790
Title: Endoscopic Ultrasound Guided Liver Biopsy Using a 19-gauge Fine Needle Biopsy Needle
Brief Title: Liver Biopsy Using a 19 Gauge Fine Needle Biopsy Needle
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A competing study made it challenging to enroll subjects.
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1354057
Record Dates: First submitted 2019-03-25; First posted 2019-04-10 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Liver Biopsy
Keywords: livery biopsy; fine needle biopsy; 19-gauge needle

STUDY DESIGN:
Intervention Model Description: This research will be carried out in a non-randomized, prospective trial pattern.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 19 Gauge needle liver biopsy (Experimental): Obtaining liver tissue with a 19 gauge core needle
  Interventions: Device: 19 gauge needle liver biopsy

INTERVENTIONS:
Device: 19 gauge needle liver biopsy — Obtaining liver tissue with a 19 gauge core needle and whether a good core biopsy can be obtained without the use of suction and secondly to determine the diagnostic yield and safety of 19 gauge core needle for liver biopsy.

SUMMARY:
A 19 gauge FNB needle, using same technique as with 22 gauge needle, to obtain liver histological specimen in regards to core length and the number of Complete Portal Triads.

DETAILED DESCRIPTION:
Liver biopsy (LB) has historically been performed by percutaneous route without image guidance (blind biopsy). However, in the last several years there has been more reliance on image guidance ultrasound-guided (USG) or computed tomography (CT) to direct the needle into the liver with the hope of limiting complications 1. Other ways of performing liver biopsy are transjugular fluoroscopy guided approach when percutaneous route is deemed not safe because of coagulopathy or ascites 2. Surgical LB (either laparoscopic or open) is yet another way of obtaining liver tissue.

Endoscopic ultrasound guided liver biopsy (EUS-LB) is proposed as a newer method that may offer several potential advantages over existing techniques for attaining liver tissue 3-8. It can be performed in an outpatient setting and offers the comfort of sedation and analgesia. EUS-LB is a technically reproducible approach regardless of body habitus, because the needle only requires traversing the gastric or duodenal wall to reach hepatic parenchyma. It also offers the benefit of a comprehensive evaluation of the GI tract, including screening or surveying for esophageal varices. EUS provides high resolution images of left lobe of the liver and a good portion of the right lobe of the liver. This coupled with Doppler capability the biopsy needle can be safely directed into the liver for sampling under real time image guidance. Intervening structures such as pleura, bowel loops and gallbladder can be easily seen by EUS and thus avoided that further decreases the risk of adverse events. It has been recognized that sampling error can lead to diagnostic inaccuracy of a biopsy from a single site 9. As compared to USG or CT scan the EUS allows easy and safe biopsy of both left and right lobes of the liver during same setting, potentially addressing concerns about sampling error.

The cost of the endoscopic procedure is the main expense of EUS-LB. Thus, this approach is best used for patients requiring EUS for evaluation of elevated liver tests. If no obstructive lesion is identified by EUS that will require ERCP then it would cost-effective to perform EUS LB during the same setting without much additional time and risks. This approach can spare the patient the additional discomfort and expense of a second dedicated LB procedure by any of the other available techniques (percutaneous, transjugular etc.). In such setting the equipment costs for the EUS-LB will mainly include only the Fine Needle Biopsy (FNB) needle, which is similar in expense to the cost of needles for the transjugular or percutaneous approach.

The traditionally used transcutaneous LB needle is 16 gauge (G) while largest EUS biopsy needle is 19 gauge. The smaller size of the needle is expected to decrease the complications rate (mainly pain and bleeding) even further. Many studies using a 19 gauge Tru-cut biopsy or Fine Needle Aspiration (FNA) needle to acquire liver tissue have obtained specimens adequate for histologic diagnosis 3-7 but there has been a wide range of specimen adequacy (19-100%). Overall, there is limited data comparing the diagnostic yield of different FNA and FNB needles.

In a recently reported systematic review and meta-analysis 10, the insufficient specimen rate with 19 gauge FNA needle was 4% compared with 20% with 19 gauge core needles, with a p value of 0.03. FNA needle demonstrated a non-significant trend toward better diagnostic results (95.8% vs 92.7%, p=0.59) and a non-significant trend toward lower rates of adverse-events (0.9% vs 2.7%, p=0.28) when compared with the core biopsy needles. The 19-gauge FNA needle used was EchoTip (Wilson Cook Medical) in one study 6 and Expect (Boston Scientific) in rest two studies 8,11. The various types of core needles used were Quick-Core 12, Pro-Core 12, SharkCore 13,14, and the Acquire needle 15.

The 19 gauge FNA needle was used in 22 patients and yielded adequate tissue for histological analysis in 20 (91 %) of them 6. In the largest multi-center EUS-LB study of 110 patients 8 where a 19 gauge FNA needle was used for liver biopsy, bilobular liver biopsy was obtained in 68 patients (62%). Even though 108 (98 %) of 110 patients yielded specimens sufficient for definitive pathological diagnosis, there were five patients where the tissue yield was less than 6 complete portal triads (CPTs) with aggregate length less than 15 mm; the value used as a reference standard in recent studies 4-6. The rate of complications was very low (1/110) 0.9% in this study.

Two ex-vivo studies demonstrated the significantly superior histologic yield, with a greater number of CPT, obtained using the novel 19 gauge SharkCore FNB 16 and 22 gauge SharkCore FNB needles 16,17, compared with 18 gauge percutaneous needles and existing 19 gauge FNA and other core needles.

The study team prospectively aimed at evaluating the diagnostic adequacy and safety of EUS-LB using a 22 gauge FNB needle while using proper technique of tissue expression from the needle to prevent fragmentation of the specimen. Forty patients underwent EUS-LB. Adequate core tissue for histopathological evaluation was obtained in all 40 patients (100%) without the use of suction. The overall tissue yield per pass was a median core length (longest fragment per pass) of 5 mm (range 2mm-33mm) and median CPT of 17 (range 8-65). The most common minor complication was mild abdominal pain in 3 patients (17.6 %) at 24 hours. There were no major complications, and no immediate or delayed bleeding (presented at DDW 2018).

In this study the study team will use a 19 gauge FNB needle, using same technique as with 22 gauge needle, to obtain liver histological specimen in regards to core length and the number of CPT.

ELIGIBILITY:
Inclusion Criteria:

1. All patients referred to Florida Hospital Endoscopy Unit for assessment of elevated liver tests with EUS and are found to have no obstructive lesion to explain elevation of liver tests and will not require ERCP.
2. Age ≥ 19 years
3. Willing to provide informed consent verbal or written.

Exclusion Criteria:

1. Age <19 years
2. Unable to safely undergo EUS for any reason
3. Coagulopathy (INR >1.6, Thrombocytopenia with platelet count <50,000/ml) for subjects on anti-coagulation therapy.
4. Unwilling or cognitively unable to provide informed consent verbal or written.
5. Pregnancy (confirmed with Standard of Care urine pregnancy test for all women with child-bearing potential only)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Diagnostic adequacy | At time of procedure
  Determine the diagnostic adequacy of the liver biopsy specimen by obtaining a histological specimen using a smaller (19 G) caliber needle. Diagnostic adequacy is defined as a sample that provides definitive pathological diagnosis (yes, no).

SECONDARY OUTCOMES:
Technique | At time of procedure
  Refine and determine the optimal technique of EUS-LB determined by the diagnostic adequacy of the liver biopsy specimen
Suction | At time of procedure
  Sample was obtained using suction (yes/no).
Number of passes | At time of procedure
  Assessing the median number of passes required to obtain diagnostically adequate histological samples histological samples histological samples
Needle Dysfunction | At time of procedure
  Did needle dysfunction occur (yes/no)?
Technical failure | At time of procedure
  Was there a technical failure (yes/no)?
Complications/Bleeding | At time of procedure; 3 days post-procedure; & 30 days post procedure
  Assessing subjects for post-procedural complications via follow up phone calls. Bleeding (yes/no).
Complications/Pain | At time of procedure; 3 days post-procedure; & 30 days post procedure
  Assessing subjects for post-procedural complications via follow up phone calls. Pain (yes/no).
Complications/Infection | At time of procedure; 3 days post-procedure; & 30 days post procedure
  Assessing subjects for post-procedural complications via follow up phone calls. Infection (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan, MD, Principal Investigator — Florida Hospital (AdventHealth Orlando)
Locations (1):
- Center for Interventional Endoscopy - Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data.

REFERENCES:
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014
- [Background] Kalambokis G, Manousou P, Vibhakorn S, Marelli L, Cholongitas E, Senzolo M, Patch D, Burroughs AK. Transjugular liver biopsy--indications, adequacy, quality of specimens, and complications--a systematic review. J Hepatol. 2007 Aug;47(2):284-94. doi: 10.1016/j.jhep.2007.05.001. Epub 2007 May 24. PMID 17561303
- [Background] Mathew A. EUS-guided routine liver biopsy in selected patients. Am J Gastroenterol. 2007 Oct;102(10):2354-5. doi: 10.1111/j.1572-0241.2007.01353_7.x. No abstract available. PMID 17897349
- [Background] Gleeson FC, Clayton AC, Zhang L, Clain JE, Gores GJ, Rajan E, Smyrk TC, Topazian MD, Wang KK, Wiersema MJ, Levy MJ. Adequacy of endoscopic ultrasound core needle biopsy specimen of nonmalignant hepatic parenchymal disease. Clin Gastroenterol Hepatol. 2008 Dec;6(12):1437-40. doi: 10.1016/j.cgh.2008.07.015. Epub 2008 Jul 26. PMID 19081532
- [Background] Dewitt J, McGreevy K, Cummings O, Sherman S, Leblanc JK, McHenry L, Al-Haddad M, Chalasani N. Initial experience with EUS-guided Tru-cut biopsy of benign liver disease. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):535-42. doi: 10.1016/j.gie.2008.09.056. PMID 19231495
- [Background] Stavropoulos SN, Im GY, Jlayer Z, Harris MD, Pitea TC, Turi GK, Malet PF, Friedel DM, Grendell JH. High yield of same-session EUS-guided liver biopsy by 19-gauge FNA needle in patients undergoing EUS to exclude biliary obstruction. Gastrointest Endosc. 2012 Feb;75(2):310-8. doi: 10.1016/j.gie.2011.09.043. PMID 22248599
- [Background] Nakai Y, Samarasena JB, Iwashita T, Park DH, Lee JG, Hu KQ, Chang KJ. Autoimmune hepatitis diagnosed by endoscopic ultrasound-guided liver biopsy using a new 19-gauge histology needle. Endoscopy. 2012;44 Suppl 2 UCTN:E67-8. doi: 10.1055/s-0031-1291567. Epub 2012 Mar 6. No abstract available. PMID 22396285
- [Background] Diehl DL, Johal AS, Khara HS, Stavropoulos SN, Al-Haddad M, Ramesh J, Varadarajulu S, Aslanian H, Gordon SR, Shieh FK, Pineda-Bonilla JJ, Dunkelberger T, Gondim DD, Chen EZ. Endoscopic ultrasound-guided liver biopsy: a multicenter experience. Endosc Int Open. 2015 Jun;3(3):E210-5. doi: 10.1055/s-0034-1391412. Epub 2015 Feb 27. PMID 26171433
- [Background] Maharaj B, Maharaj RJ, Leary WP, Cooppan RM, Naran AD, Pirie D, Pudifin DJ. Sampling variability and its influence on the diagnostic yield of percutaneous needle biopsy of the liver. Lancet. 1986 Mar 8;1(8480):523-5. doi: 10.1016/s0140-6736(86)90883-4. PMID 2869260
- [Background] Mohan BP, Shakhatreh M, Garg R, Ponnada S, Adler DG. Efficacy and safety of EUS-guided liver biopsy: a systematic review and meta-analysis. Gastrointest Endosc. 2019 Feb;89(2):238-246.e3. doi: 10.1016/j.gie.2018.10.018. Epub 2018 Oct 31. PMID 30389469
- [Background] Gor N, Salem SB, Jakate S, Patel R, Shah N, Patil A. Histological adequacy of EUS-guided liver biopsy when using a 19-gauge non-Tru-Cut FNA needle. Gastrointest Endosc. 2014 Jan;79(1):170-2. doi: 10.1016/j.gie.2013.06.031. Epub 2013 Jul 31. No abstract available. PMID 23916397
- [Background] Sey MS, Al-Haddad M, Imperiale TF, McGreevy K, Lin J, DeWitt JM. EUS-guided liver biopsy for parenchymal disease: a comparison of diagnostic yield between two core biopsy needles. Gastrointest Endosc. 2016 Feb;83(2):347-52. doi: 10.1016/j.gie.2015.08.012. Epub 2015 Aug 13. PMID 26278654
- [Background] Nieto J, Khaleel H, Challita Y, Jimenez M, Baron TH, Walters L, Hathaway K, Patel K, Lankarani A, Herman M, Holloman D, Saab S. EUS-guided fine-needle core liver biopsy sampling using a novel 19-gauge needle with modified 1-pass, 1 actuation wet suction technique. Gastrointest Endosc. 2018 Feb;87(2):469-475. doi: 10.1016/j.gie.2017.05.013. Epub 2017 May 24. PMID 28551024
- [Background] Shah ND, Sasatomi E, Baron TH. Endoscopic Ultrasound-guided Parenchymal Liver Biopsy: Single Center Experience of a New Dedicated Core Needle. Clin Gastroenterol Hepatol. 2017 May;15(5):784-786. doi: 10.1016/j.cgh.2017.01.011. Epub 2017 Jan 23. No abstract available. PMID 28126424
- [Background] Lee WJ, Uradomo LT, Zhang Y, Twaddell W, Darwin P. Comparison of the Diagnostic Yield of EUS Needles for Liver Biopsy: Ex Vivo Study. Diagn Ther Endosc. 2017;2017:1497831. doi: 10.1155/2017/1497831. Epub 2017 Sep 13. PMID 29056843
- [Background] Schulman AR, Thompson CC, Odze R, Chan WW, Ryou M. Optimizing EUS-guided liver biopsy sampling: comprehensive assessment of needle types and tissue acquisition techniques. Gastrointest Endosc. 2017 Feb;85(2):419-426. doi: 10.1016/j.gie.2016.07.065. Epub 2016 Aug 13. PMID 27530070
- [Background] Rombaoa C CA. Mo1351 The safety and feasibileity of endoscopic ultrasound-guided parenchymal liver biopsy at a large community hospital. Gastrointestinal endoscopy; 87(6): AB458.